CLINICAL TRIAL: NCT05928403
Title: Rate of Return to Sport After Total Knee Prosthesis: Comparison of Three Different Types of Prostheses (Medial Pivot, Medial Bearing and Cruciate Retaining)
Brief Title: Rate of Return to Sport After Total Knee Prosthesis: Comparison of Three Types of Prostheses
Acronym: TKA&RTS
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00626-39
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- medial pivot: Return to sport rate for patients with a Medial Pivot knee prosthesis
  Interventions: Other: total knee prosthesis
- medial bearing: Return to sport rate for patients with a Medial Bearing knee prosthesis
  Interventions: Other: total knee prosthesis
- cruciate retaining: Return to sport rate for patients with a Cruciate Retaining prosthesis
  Interventions: Other: total knee prosthesis

INTERVENTIONS:
Other: total knee prosthesis — Comparison of three cohorts on the return to sport of patients after total knee prosthesis according to the type of prosthesis

SUMMARY:
The purpose of the study is the rate of return to sport (regardless of the sport envisaged) after a minimum of 3 years after total knee prosthesis.

DETAILED DESCRIPTION:
This is an ambispective, comparative study of three cohorts, non-randomized, open, monocentric, relating to the return to sport of patients who have benefited from one of the three designs of prostheses under study (medial pivot, medial bearing and cruciate retaining) after total knee prosthesis.

Patients who received a total knee prosthesis with medial pivot, medial bearing and cruciate retaining prosthesis between 2018 and 2020 will be called by the investigator, and the study will be offered to them (D-3 to D0). The investigator will explain the study to the patient, send him the information note electronically and answer all his questions about the study. If the patient agrees to participate after a reflection period, the inclusion (D0) will be documented in the medical file, and the patient will be assessed the same day by telephone using the assessments set up in the study, except for the questionnaires on his functional and physical abilities that will be sent to him electronically. The patient will return his answers to the questionnaires on this same email address or by telephone according to his preference. A secure and unique email address will be created by the principal investigator for the purposes of the study and for use strictly specific to the study, in the investigating center.

ELIGIBILITY:
Inclusion Criteria:

* First total knee prosthesis between 2018 and 2020;
* Conventional alignment technique using the same surgical technique for total knee prosthesis;
* Placement of a medial pivot prosthesis (Evolution®), mobile bearing (SCORE® Amplitude) or traditional cruciate retaining prosthesis (Stryker® Triathlon);
* Affiliation to a social security scheme;
* Patient having been informed and having given his oral non-objection

Exclusion Criteria:

* Bilateral total knee prosthesis;
* Medical history of revision of Total Knee Prosthesis;
* Articulation malformation of the lower limbs;
* Having undergone revision surgery;
* Inability to understand information related to the study for linguistic, psychological, cognitive reasons;
* Patient under legal protection, or deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible on retrospective criteria. These are patients who underwent total knee prosthesis surgery between 2018 and 2020 with placement of a medial pivot, medial bearing and cruciate retaining type prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
rate of return to sport | 3 years
  rate of return to sport after a minimum of 3 years after total knee prosthesis

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Aguiléra, Biarritz
  - Clinique des Cèdres, Cornebarrieu

IPD SHARING:
Plan to Share IPD: No